CLINICAL TRIAL: NCT00745108
Title: A Multinational, Multicenter, Randomized, Double-blind, Parallel Group, Active Controlled, Comparative Trial, to Assess the Endometrial Histological Profile Following Treatment With Tibolone (Org OD14) Versus Conjugated Estrogen (CE) Plus Medroxyprogesterone Acetate (MPA) in Postmenopausal Women
Brief Title: Tibolone Endometrium Study (Study 32972)(P06470)
Acronym: THEBES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P06470; 32972
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Postmenopausal Women
MeSH Terms: interventions — tibolone; N-(2-chloroethyl)-N-methylphenylalanine; Estrogens, Conjugated (USP); Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tibolone 1.25 mg (Experimental)
  Interventions: Drug: tibolone
- Tibolone 2.5 mg (Experimental)
  Interventions: Drug: Tibolone 2.5 mg
- CE/MPA (Active Comparator)
  Interventions: Drug: CE/MPA

INTERVENTIONS:
Drug: tibolone — oral 1.25 mg tablet, once daily, for 2 years
  Arms: Tibolone 1.25 mg
Drug: Tibolone 2.5 mg — oral 2.5 mg tablet, once daily, for 2 years
  Other Names: Livial
  Arms: Tibolone 2.5 mg
Drug: CE/MPA — oral, 0.625 mg tablet conjugated equine estrogen and 2.5 mg medroxyprogesterone acetate tablet placed together in a single capsule, once daily, for 2 years
  Other Names: Premarin; Provera
  Arms: CE/MPA

SUMMARY:
Tibolone has been registered for the treatment of climacteric symptoms and for the prevention of postmenopausal osteoporosis. This is a 2-year study to further confirm the endometrial safety of tibolone in comparison with CE/MPA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women, 45 to 65 years of age with an intact uterus. Women must have been postmenopausal for less than 15 years, have an atrophic or inactive endometrium, and a body mass index of 18 - 32 kg/ m2 (inclusive).

Exclusion Criteria:

* Final diagnosis of the endometrial biopsy as 'no tissue' or 'tissue insufficient for diagnosis'.
* Double layer endometrial thickness > 6 mm as assessed by transvaginal ultrasonography (TVUS).
* Any previous or current unopposed estrogen administration or tamoxifen citrate.
* Any unexplained vaginal bleeding following the menopause.
* Women with abnormal Pap smear test results (PAP IIb and higher)
* Previous use of raloxifene hydrochloride for longer than one month.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2001-10-01 (Actual); Primary Completion 2005-07-21 (Actual); Study Completion 2005-07-21 (Actual)

PRIMARY OUTCOMES:
Endometrial biopsy and histological examination | At 1 year and 2 year.

SECONDARY OUTCOMES:
Double-layer endometrial thickness by transvaginal ultrasonography (TVUS), vaginal bleeding from a Bleeding Episode Log. | TVUS: at 1 year and 2 year; Vaginal bleeding: daily recording

REFERENCES:
- [Background] Archer DF, Hendrix S, Ferenczy A, Felix J, Gallagher JC, Rymer J, Skouby SO, den Hollander W, Stathopoulos V, Helmond FA; THEBES Study Group. Tibolone histology of the endometrium and breast endpoints study: design of the trial and endometrial histology at baseline in postmenopausal women. Fertil Steril. 2007 Oct;88(4):866-78. doi: 10.1016/j.fertnstert.2006.12.052. Epub 2007 Jun 4. PMID 17548089